CLINICAL TRIAL: NCT06087133
Title: Prenatal Starting Early Program: Randomized Controlled Trial of an mHealth Intervention in Prenatal Care and Wic to Improve Nutrition and Physical Activity During Pregnancy
Brief Title: Prenatal Starting Early Program mHealth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-00902
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy
Keywords: Prenatal care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Care + StEP:Prenatal (Experimental): Participants will receive routine care and up to 8 StEP:Prenatal sessions. Routine care will follow through the post-partum period.
  Interventions: Behavioral: StEP:Prenatal; Other: Routine Care
- Routine Care (Active Comparator): Participants will receive routine care during pregnancy and the post-partum period.
  Interventions: Other: Routine Care

INTERVENTIONS:
Behavioral: StEP:Prenatal — StEP is a health care-based intervention based on elements of Social Cognitive Theory, in which registered dietitians with additional certified lactation counselor training (RD/CLC) provide individual and group-based support for healthy diet, physical activity, other lifestyle behaviors, stress reduction, and healthy gestational weight gain. StEP:Prenatal will be delivered remotely. There are up to 8 sessions scheduled around the routine prenatal care visits and designed to be offered from the first trimester of pregnancy through delivery.
  Arms: Routine Care + StEP:Prenatal
Other: Routine Care — Routine care includes routine prenatal and post-partum primary care visits, on-site WIC services and referrals for additional services as needed (e.g., women with poor weight gain, obesity, or diabetes may be offered additional nutrition visits).

SUMMARY:
The purpose of this interventional trial is to test the efficacy of the remote delivery of the StEP:Prenatal intervention compared to standard prenatal care in pregnant individuals planning to receive prenatal and pediatric care at Bellevue Hospital. The primary aims are to determine the efficacy of the remotely delivered StEP:Prenatal intervention on diet, lifestyle behaviors, social determinants of health (SDoH), and pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant in the first trimester (up to 13 weeks, 6 days)
* Speak English or Spanish fluently
* Intent to receive prenatal and pediatric care at Bellevue
* ≥18 years
* Have a smart phone or device with internet access
* Willing and able to provide consent

Exclusion Criteria:

* Severe illness (severe medical or mental health condition e.g. cancer, epilepsy neuromuscular disease, psychosis or bipolar disorder).

Note: Diabetes, hypertension, depression are not excluded.

* Living in a shelter
* Receiving treatment for drug or alcohol use

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Daily servings of fruits (cup equivalents) | Week 28-42 (third trimester)
  As Measured by the Diet History Questionnaire (DHQ) III. The DHQ III consists of 135 food and beverage line items and 26 dietary supplement questions.
  Self-reported by each participant via DHQ III.
Daily servings of whole grains (ounce equivalents) | Week 28-42 (third trimester)
  As Measured by the Diet History Questionnaire (DHQ) III. The DHQ III consists of 135 food and beverage line items and 26 dietary supplement questions.
  Self-reported by each participant via DHQ III.
Daily servings of refined grains (ounce equivalents) | Week 28-42 (third trimester)
  As Measured by the Diet History Questionnaire (DHQ) III. The DHQ III consists of 135 food and beverage line items and 26 dietary supplement questions.
  Self-reported by each participant via DHQ III.
Daily servings of dairy (total milk cup equivalents) | Week 28-42 (third trimester)
  As Measured by the Diet History Questionnaire (DHQ) III. The DHQ III consists of 135 food and beverage line items and 26 dietary supplement questions.
  Self-reported by each participant via DHQ III.
Daily servings of vegetables (cup equivalents) | Week 28-42 (third trimester)
  As Measured by the Diet History Questionnaire (DHQ) III. The DHQ III consists of 135 food and beverage line items and 26 dietary supplement questions.
  Self-reported by each participant via DHQ III.
Number of times 100% pure fruit juice consumed | Week 28-42 (third trimester)
  Self-reported using survey items from the Behavioral Risk Factor Surveillance System (BRFSS).
  The question is related to 100% fruit juice consumed during the past 30 days.
Number of times sugar sweetened beverages (not including 100% fruit juice) consumed | Week 28-42 (third trimester)
  Self-reported using survey items from the Behavioral Risk Factor Surveillance System (BRFSS).
  The questions are related to sugar sweetened beverages (not including 100% fruit juice) consumed during the past 30 days.
Daily servings of protein foods (ounce equivalents) | Week 28-42 (third trimester)
  As Measured by the Diet History Questionnaire (DHQ) III. The DHQ III consists of 135 food and beverage line items and 26 dietary supplement questions.
  Self-reported by each participant via DHQ III.
Healthy Eating Index (HEI)-2015 score | Week 28-42 (third trimester)
  The HEI-2015 measures 13 components (9 adequacy [total fruits, whole fruits, total vegetables, greens and beans, whole grains, dairy, total protein foods, seafood and plant proteins, fatty acids], and 4 moderation [refined grains, sodium, saturated fat, added sugars]. For the adequacy components, higher scores indicate higher intakes. For the moderation components, higher scores reflect lower intakes. Scores for each component are summed to create a total maximum HEI-2020 score of 100 points, with a higher score reflecting a dietary pattern that better aligns with the dietary guidelines.
  HEI scores range from 0 to 100, with higher scores indicating better diet quality. HEI scores > 80 indicate a "good" diet, scores ranging from 51 to 80 reflect a diet that "needs improvement," and HEI scores < 51 imply a "poor" diet (7).
Daily servings of fruits (cup equivalents) | 3 months (6-14 weeks postpartum)
  As Measured by the Diet History Questionnaire (DHQ) III. The DHQ III consists of 135 food and beverage line items and 26 dietary supplement questions.
  Self-reported by each participant via DHQ III.
Daily servings of whole grains (ounce equivalents) | 3 months (6-14 weeks postpartum)
  As Measured by the Diet History Questionnaire (DHQ) III. The DHQ III consists of 135 food and beverage line items and 26 dietary supplement questions.
  Self-reported by each participant via DHQ III.
Daily servings of refined grains (ounce equivalents) | 3 months (6-14 weeks postpartum)
  As Measured by the Diet History Questionnaire (DHQ) III. The DHQ III consists of 135 food and beverage line items and 26 dietary supplement questions.
  Self-reported by each participant via DHQ III.
Daily servings of dairy (total milk cup equivalents) | 3 months (6-14 weeks postpartum)
  As Measured by the Diet History Questionnaire (DHQ) III. The DHQ III consists of 135 food and beverage line items and 26 dietary supplement questions.
  Self-reported by each participant via DHQ III.
Daily servings of vegetables (cup equivalents) | 3 months (6-14 weeks postpartum)
  As Measured by the Diet History Questionnaire (DHQ) III. The DHQ III consists of 135 food and beverage line items and 26 dietary supplement questions.
  Self-reported by each participant via DHQ III.
Daily servings of protein foods (ounce equivalents) | 3 months (6-14 weeks postpartum)
  As Measured by the Diet History Questionnaire (DHQ) III. The DHQ III consists of 135 food and beverage line items and 26 dietary supplement questions.
  Self-reported by each participant via DHQ III.
Number of times 100% pure fruit juice consumed | 3 months (6-14 weeks postpartum)
  Self-reported using survey items from the Behavioral Risk Factor Surveillance System (BRFSS).
  The question is related to 100% fruit juice consumed during the past 30 days.
Number of times sugar sweetened beverages (not including 100% fruit juice) consumed | 3 months (6-14 weeks postpartum)
  Self-reported using survey items from the Behavioral Risk Factor Surveillance System (BRFSS).
  The questions are related to sugar sweetened beverages (not including 100% fruit juice) consumed during the past 30 days.
Healthy Eating Index (HEI)-2015 score | 3 months (6-14 weeks postpartum)
  The HEI-2015 measures 13 components (9 adequacy [total fruits, whole fruits, total vegetables, greens and beans, whole grains, dairy, total protein foods, seafood and plant proteins, fatty acids], and 4 moderation [refined grains, sodium, saturated fat, added sugars]. For the adequacy components, higher scores indicate higher intakes. For the moderation components, higher scores reflect lower intakes. Scores for each component are summed to create a total maximum HEI-2020 score of 100 points, with a higher score reflecting a dietary pattern that better aligns with the dietary guidelines.
  HEI scores range from 0 to 100, with higher scores indicating better diet quality. HEI scores > 80 indicate a "good" diet, scores ranging from 51 to 80 reflect a diet that "needs improvement," and HEI scores < 51 imply a "poor" diet (7).
Total amount of screen time | Week 28-42 (third trimester)
  Self-reported using survey items from the Behavioral Risk Factor Surveillance System (BRFSS).
  The questions are related to daily activities, physical activities, and sedentary activities.
Total amount of physical activity | Week 28-42 (third trimester)
  Self-reported using survey items from the Behavioral Risk Factor Surveillance System (BRFSS).
  The questions are related to daily activities, physical activities, and sedentary activities.
Total amount of screen time | 3 months (6-14 weeks postpartum)
  Self-reported using survey items from the Behavioral Risk Factor Surveillance System (BRFSS).
  The questions are related to daily activities, physical activities, and sedentary activities.
Total amount of physical activity | 3 months (6-14 weeks postpartum)
  Self-reported using survey items from the Behavioral Risk Factor Surveillance System (BRFSS).
  The questions are related to daily activities, physical activities, and sedentary activities.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) score | Week 28-42 (third trimester)
  Patient Health Questionnaire-9 (PHQ-9) measures depressive symptoms and consists of 9 items.
  The PHQ-9 total score ranges from 0 to 27 (scores of 5-9 are classified as mild depressive symptoms; 10-14 as moderate depressive symptoms; 15-19 as moderately severe depressive symptoms; ≥ 20 as severe depressive symptoms).
Patient Health Questionnaire (PHQ-9) score | 3 months (6-14 weeks postpartum)
  Patient Health Questionnaire-9 (PHQ-9) measures depressive symptoms and consists of 9 items.
  The PHQ-9 total score ranges from 0 to 27 (scores of 5-9 are classified as mild depressive symptoms; 10-14 as moderate depressive symptoms; 15-19 as moderately severe depressive symptoms; ≥ 20 as severe depressive symptoms).
Generalized Anxiety Disorder-7 score | Week 28-42 (third trimester)
  Generalized Anxiety Disorder-7 score (GAD-7) measures anxiety symptoms and consists of 7 items.
  The GAD-7 total score ranges from 0 to 21 (scores of 0-4 are classified as minimal anxiety symptoms; 5-9 as mild anxiety symptoms; 10-14 as moderate anxiety symptoms; 15-21 as severe anxiety symptoms).
Generalized Anxiety Disorder-7 score | 3 months (6-14 weeks postpartum)
  Generalized Anxiety Disorder-7 score (GAD-7) measures anxiety symptoms and consists of 7 items.
  The GAD-7 total score ranges from 0 to 21 (scores of 0-4 are classified as minimal anxiety symptoms; 5-9 as mild anxiety symptoms; 10-14 as moderate anxiety symptoms; 15-21 as severe anxiety symptoms).
Perceived Stress Scale score | Week 28-42 (third trimester)
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Perceived Stress Scale score | 3 months (6-14 weeks postpartum)
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Family Resilience score | Week 28-42 (third trimester)
  An overall family resilience score is calculated using the mean from each of the participants' responses to the 4 items. Scores range from 0 to 4. Higher scores indicate greater family resilience.
Family Resilience score | 3 months (6-14 weeks postpartum)
  An overall family resilience score is calculated using the mean from each of the participants' responses to the 4 items. Scores range from 0 to 4. Higher scores indicate greater family resilience.
Gestational weight gain | 3 months (6-14 weeks postpartum)
Total number of remote StEP:Prenatal sessions attended | 3 months (6-14 weeks postpartum)
Total number of pregnancy care visits attended | 3 months (6-14 weeks postpartum)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Messito, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYC Health + Hospitals/Bellevue, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Mary.Messito@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Mary.Messito@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT06087133/ICF_000.pdf